CLINICAL TRIAL: NCT05365191
Title: Development and Utilization of Indocyanine Green Fluorescence Near Infrared Zone II Lymphography in Breast Cancer Patients
Brief Title: A Study Evaluating Near-infrared Zone II Imaging in Sentinel Lymph Node Mapping in Breast Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital Hsin-Chu Branch (Other)
Collaborators: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 110-163-F
Record Dates: First submitted 2022-04-27; First posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Breast Cancer; Sentinel Lymph Node
Keywords: Indocyanine green; Image-guided surgery; Multispectral fluorescence imaging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: The participants will be assigned to one single arm that accepted both near infrared zone I and near infrared zone II imaging during the near infrared fluorescence navigated sentinel lymph node biopsy procedure.
Masking Description: The patient will know they are going to accept near infrared zone II imaging during the sentinel lymph node biopsy procedure. They will not see the images and will not know the quality results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multispectral near infrared imaging (Other): The participants will be assigned to one single arm that accepted both near infrared zone I and near infrared zone II imaging during the near infrared fluorescence navigated sentinel lymph node biopsy procedure. Imaging quality will be compared between different spectrums.
  Interventions: Procedure: Near infrared fluorescence navigated sentinel lymph node mapping

INTERVENTIONS:
Procedure: Near infrared fluorescence navigated sentinel lymph node mapping — Participants undergo sentinel lymph node biopsy for breast cancer, and use blue dye/Tc99m radioisotope as primary tracer. Indocyanine green near infrared fluorescence as secondary tracer for mapping.

SUMMARY:
This study aims for evaluating near infrared zone II imaging in sentinel lymph node mapping in breast cancer patients.

DETAILED DESCRIPTION:
Multi-wavelength fluorescence has been surveyed in various fields of surgery. However, it was still under investigation, and has not been matured for clinical use. This study will evaluate near infrared zone II spectrums for breast cancer patient undergoing sentinel lymph node mapping with near-infrared fluorescence navigation.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer, adults

Exclusion Criteria:

* Patient aged < 20 years old
* Primary lesion without indication of sentinel lymph node biopsy in current guidelines (Low-risk ductal carcinoma in situ or metastatic breast cancer)
* Patient who is allergic to primary tracers (including Tc99m and blue dye)
* Patient who is allergic to indocyanine green

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04-08 (Actual); Primary Completion 2023-04-07 (Estimated); Study Completion 2023-04-07 (Estimated)

PRIMARY OUTCOMES:
Signal-to-background ratio (SBR) | through study completion, an average of 1 year
  Evaluates the SBR of the near-infrared fluorescence between the retrieved sentinel lymph nodes and the background.

SECONDARY OUTCOMES:
Sentinel lymph nodes pathology | through study completion, an average of 1 year
  The positivity and number of retrieved sentinel lymph nodes at definitive pathology report.
Penetration depth | through study completion, an average of 1 year
  Evaluates the depth of the deepest visualized subcutaneous lymphatics in the breast

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Chun Hsieh, MD, Study Chair — National Taiwan University Hospital Hsin-Chu Branch
Locations (1):
- National Taiwan University Hospital Hsin-Chu Branch Biomedical Park Hospital, Zhubei, HsinChu County, Taiwan

REFERENCES:
- [Background] Hu Z, Fang C, Li B, Zhang Z, Cao C, Cai M, Su S, Sun X, Shi X, Li C, Zhou T, Zhang Y, Chi C, He P, Xia X, Chen Y, Gambhir SS, Cheng Z, Tian J. First-in-human liver-tumour surgery guided by multispectral fluorescence imaging in the visible and near-infrared-I/II windows. Nat Biomed Eng. 2020 Mar;4(3):259-271. doi: 10.1038/s41551-019-0494-0. Epub 2019 Dec 23. PMID 31873212
- [Background] van Beurden F, van Willigen DM, Vojnovic B, van Oosterom MN, Brouwer OR, der Poel HGV, Kobayashi H, van Leeuwen FWB, Buckle T. Multi-Wavelength Fluorescence in Image-Guided Surgery, Clinical Feasibility and Future Perspectives. Mol Imaging. 2020 Jan-Dec;19:1536012120962333. doi: 10.1177/1536012120962333. PMID 33125289